CLINICAL TRIAL: NCT00096824
Title: International Neurological Study: A Stand Alone Study for Participants of A5175 (A Phase IV, Randomized, Open-Label Evaluation of the Efficacy of Once-Daily Protease Inhibitor and Once-Daily Non-Nucleoside Reverse Transcriptase Inhibitor-Containing Therapy Combination for Initial Treatment of HIV-1 Infected Individuals From Diverse Areas of the World)
Brief Title: A Study of Dementia and Neurological Problems in HIV Infected Patients Who Are Participating in ACTG A5175
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5199; 1U01AI068636 (NIH)
Record Dates: First submitted 2004-11-15; First posted 2004-11-16 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Participants will undergo neurological examinations and neuropsychological assessments at entry to both steps of ACTG A5175 and before the administration of the new antiretroviral regimen, then every 24 weeks until they discontinue ACTG A5175. Physicians will make targeted diagnoses at each study visit.
  Interventions: Behavioral: Neurological assessment

INTERVENTIONS:
Behavioral: Neurological assessment — All participants will undergo neurological examinations and neuropsychological assessments.

SUMMARY:
The purpose of this study is to determine how often dementia and other neurological problems occur in people with HIV. Participants of ACTG A5175 will enroll in this study.

DETAILED DESCRIPTION:
Both the central and peripheral nervous systems (CNS and PNS) are affected by HIV; however, the causes of neurotoxicity in HIV infected patients are unknown. Initial data indicate that as many as 40% of patients with HIV develop some form of dementia. Other common neurological problems observed in HIV patients are peripheral neuropathy and opportunistic infections of the CNS. Most antiretroviral drugs used in the treatment of HIV have poor penetration into the CNS, which may explain how HIV persists in the CNS and contributes to the prevalence of dementia and other neurological disorders in HIV infected patients. This study will examine the prevalence of dementia and other neurological disorders in participants in ACTG A5175, "Once-Daily PI/NNRTI Therapy Combinations for Treatment Naive, HIV Infected Patients in Resource-limited Conditions."

The study will last approximately 2.5 to 3 years. Participants will undergo neurological examinations and neuropsychological assessments at entry to both steps of ACTG A5175 and before the administration of the new antiretroviral regimen, then every 24 weeks until they discontinue ACTG A5175. Physicians will make targeted diagnoses at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Prior antiretroviral therapy for less than 7 days any time prior to study entry
* CD4 count less than 300 cells/mm3
* Willing to use acceptable means of contraception
* Plans to stay in the area for the duration of study participation
* Willing to adhere to study follow-up schedule for ACTG A5175 and this study
* Have not begun ACTG A5175 antiretroviral therapy, but planning to start therapy after enrolling in this study

Exclusion Criteria:

* Any active severe psychiatric illness (e.g., schizophrenia, severe depression, severe bipolar affective disorder) that, in the opinion of the site investigator, may interfere with the study results
* Current drug or alcohol abuse that, in the opinion of the site investigator, would interfere with study requirements
* Serious illness or hospitalization that, in the opinion of the site investigator, may interfere with the study results
* Any condition that, in the opinion of the site investigator, would interfere with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants who enrolled in ACTG study 5175
Sampling Method: Non-Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2006-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Robertson, PhD, Study Chair — Department of Neurology, University of North Carolina at Chapel Hill; Johnstone Kumwenda, MD, MBBS, MMED, Study Chair — Internal Medicine, Johns Hopkins Project; Khuanchai Supparatpinyo, MD, Study Chair — Research Institute for Health Sciences, Chiang Mai University
Locations (11):
- Brazil (2):
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas-Fiocruz, Rio de Janeiro
- India (4):
  - YRG Center for AIDS Research and Education, Chennai
  - Dr. Kotnis Dispensary, Pune
  - National AIDS Research Institute (NARI) ICMR, Pune
  - National Institute of Virology (NARI), Pune
- Malawi (2):
  - The Johns Hopkins-Malawi College of Medicine Project, Blantyre
  - University of North Carolina Project (UNC Project), Lilongwe
- South Africa (2):
  - University of KwaZulu Natal, Durban, KwaZulu-Natal
  - University of Witwatersrand, Johannesburg
- University of Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Background] Albright AV, Soldan SS, Gonzalez-Scarano F. Pathogenesis of human immunodeficiency virus-induced neurological disease. J Neurovirol. 2003 Apr;9(2):222-7. doi: 10.1080/13550280390194073. PMID 12707852
- [Background] McArthur JC, Haughey N, Gartner S, Conant K, Pardo C, Nath A, Sacktor N. Human immunodeficiency virus-associated dementia: an evolving disease. J Neurovirol. 2003 Apr;9(2):205-21. doi: 10.1080/13550280390194109. PMID 12707851
- [Background] Sacktor N. The epidemiology of human immunodeficiency virus-associated neurological disease in the era of highly active antiretroviral therapy. J Neurovirol. 2002 Dec;8 Suppl 2:115-21. doi: 10.1080/13550280290101094. PMID 12491162
- [Background] Sacktor N, McDermott MP, Marder K, Schifitto G, Selnes OA, McArthur JC, Stern Y, Albert S, Palumbo D, Kieburtz K, De Marcaida JA, Cohen B, Epstein L. HIV-associated cognitive impairment before and after the advent of combination therapy. J Neurovirol. 2002 Apr;8(2):136-42. doi: 10.1080/13550280290049615. PMID 11935465
- [Derived] Michael H, Rapulana A, Smit T, Xulu N, Danaviah S, Ramlall S, Oosthuizen F. Dual Trajectories of Serum Brain-Derived Neurotrophic Factor and Cognitive Function in People Living with HIV. Res Sq [Preprint]. 2025 Apr 14:rs.3.rs-4307577. doi: 10.21203/rs.3.rs-4307577/v1. PMID 40321763
- [Derived] Michael HU, Rapulana AM, Smit T, Xulu N, Danaviah S, Ramlall S, Oosthuizen F. Dual trajectories of serum brain-derived neurotrophic factor and cognitive function in people living with HIV. Sci Rep. 2025 May 3;15(1):15520. doi: 10.1038/s41598-025-99569-6. PMID 40319152
- [Derived] Robertson KR, Jiang H, Kumwenda J, Supparatpinyo K, Marra CM, Berzins B, Hakim J, Sacktor N, Campbell TB, Schouten J, Mollan K, Tripathy S, Kumarasamy N, La Rosa A, Santos B, Silva MT, Kanyama C, Firhnhaber C, Murphy R, Hall C, Marcus C, Naini L, Masih R, Hosseinipour MC, Mngqibisa R, Badal-Faesen S, Yosief S, Vecchio A, Nair A; AIDS Clinical Trials Group. Human Immunodeficiency Virus-associated Neurocognitive Impairment in Diverse Resource-limited Settings. Clin Infect Dis. 2019 May 2;68(10):1733-1738. doi: 10.1093/cid/ciy767. PMID 30219843
- [Derived] Robertson KR, Oladeji B, Jiang H, Kumwenda J, Supparatpinyo K, Campbell TB, Hakim J, Tripathy S, Hosseinipour MC, Marra CM, Kumarasamy N, Evans S, Vecchio A, La Rosa A, Santos B, Silva MT, Montano S, Kanyama C, Firnhaber C, Price R, Marcus C, Berzins B, Masih R, Lalloo U, Sanne I, Yosief S, Walawander A, Nair A, Sacktor N, Hall C; 5199 Study Team; and the AIDS Clinical Trials Group. Human Immunodeficiency Virus Type 1 and Tuberculosis Coinfection in Multinational, Resource-limited Settings: Increased Neurological Dysfunction. Clin Infect Dis. 2019 May 2;68(10):1739-1746. doi: 10.1093/cid/ciy718. PMID 30137250
- [Derived] Robertson K, Jiang H, Kumwenda J, Supparatpinyo K, Evans S, Campbell TB, Price R, Tripathy S, Kumarasamy N, La Rosa A, Santos B; 5199 study team; Silva MT, Montano S, Kanyama C, Faesen S, Murphy R, Hall C, Marra CM, Marcus C, Berzins B, Allen R, Housseinipour M, Amod F, Sanne I, Hakim J, Walawander A, Nair A; AIDS Clinical Trials Group. Improved neuropsychological and neurological functioning across three antiretroviral regimens in diverse resource-limited settings: AIDS Clinical Trials Group study a5199, the International Neurological Study. Clin Infect Dis. 2012 Sep;55(6):868-76. doi: 10.1093/cid/cis507. Epub 2012 Jun 1. PMID 22661489
- See also: Click here for more information about the ACTG A5175 study — http://clinicaltrials.gov/ct/show/NCT00084136